CLINICAL TRIAL: NCT05854004
Title: Effectiveness of Therapeutic Ultrasound and Myofascial Release Technique to Release Trigger Points to Increase Range of Motion and Pain Relief in Upper Trapezius Tightness
Brief Title: Effectiveness of TU and MRT to Release Trigger Points to Increase RoM and Pain Relief in Upper TT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/532
Record Dates: First submitted 2023-03-18; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Ultrasound (Other)
  Interventions: Diagnostic Test: Therapeutic Ultrasound
- Myofascial Release Technique (Other)
  Interventions: Diagnostic Test: Myofascial Release Technique

INTERVENTIONS:
Diagnostic Test: Therapeutic Ultrasound — Therapeutic Ultrasound to Release Trigger Points to Increase Range of Motion and Pain Relief in Upper Trapezius Tightness
  Arms: Therapeutic Ultrasound
Diagnostic Test: Myofascial Release Technique — Myofascial Release Technique to Release Trigger Points to Increase Range of Motion and Pain Relief in Upper Trapezius Tightness
  Arms: Myofascial Release Technique

SUMMARY:
To find out the Effectiveness of Therapeutic Ultrasound and Myofascial Release Technique to Release Trigger Points to Increase Range of Motion and Pain Relief in Upper Trapezius Tightness

ELIGIBILITY:
Inclusion Criteria:

* 1. Age between 20-40years.
* 2. Male and female both are included.
* 3. Those having tenderness on a taut muscle band, rise in regular pain, local twitching response, and restricted range of motion of cervical region.

Exclusion Criteria:

* 1. Those having referred pain due to any pathology of cervical.
* 2. Those having any healing fractures over upper back and in neck region.
* 3. Those who have dermatitis over upper back or any clotting disorder.
* 4. Any related wound in neck region or any pathology of shoulder.
* 5. Those who has any degenerative cervical spine disease. (2)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Numaric Pain scale Rating (NPR). | 6 Months.
  Pre and post interventions with (NPR) Scale to Increase Range of Motion and Pain Relief in Upper Trapezius Tightness

CONTACTS AND LOCATIONS:
Locations (1):
- Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No